CLINICAL TRIAL: NCT07181200
Title: Accelerating the Development of an Extended-specificity Multiplex Urine Immunoassay for the Diagnosis and Serotyping of Pneumococcal Pneumonia in High Carriage and Disease Burden Settings Like Malawi
Brief Title: Urine Pneumococcal Antigen Project
Acronym: UPAP
Status: Not yet recruiting | Type: Observational
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Malawi Liverpool Wellcome Programme (Other)
Responsible Party: Sponsor
Other Study IDs: P.0725-1685
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pneumonia; Pneumonia - Bacterial
Keywords: Urinary pneumococcal antigen; Serotype-specific urinary antigen detection
MeSH Terms: conditions — Pneumonia; Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy community: Healthy children living in Ndirande community, aged between 12 and 24 months at recruitment.
- Community pneumonia: Children aged between 12 and 24 months who have presented to Ndirande Health Centre with a pneumonia clinical syndrome (based on the WHO definition of fever, cough, tachypnoea and dyspnoea) for which they are prescribed antibiotic therapy.
- Hospital pneumonia - first admission: Children aged between 12 and 24 months who have been admitted to Queen Elizabeth Central Hospital for the first time with a pneumonia clinical syndrome (based on the WHO definition of fever, cough, tachypnoea and dyspnoea) for which they are prescribed antibiotic therapy.
- Hospital pneumonia - re-admission: Children aged between 12 and 24 months who have been re-admitted to Queen Elizabeth Central Hospital with a pneumonia clinical syndrome (based on the WHO definition of fever, cough, tachypnoea and dyspnoea) for which they are prescribed antibiotic therapy, within 3 months of a previous hospitalisation with pneumonia.

SUMMARY:
Background:Pneumonia caused by the bacteria Streptococcus pneumoniae is a leading cause of death among children under five years of age, especially in sub-Saharan Africa. Accurate diagnosis remains challenging due to the need for invasive procedures to obtain samples for culture-based diagnostic tests, which are not very sensitive for detecting S.pneumoniae, particularly after antibiotic use.

Serotype-specific urinary antigen detection (ssUAD) assays are a promising, non-invasive alternative for the surveillance and diagnosis of pneumococcal disease. Importantly, they can identify different serotypes of S.pneumoniae, which is crucial for monitoring vaccine impact. However, the ability of the ssUAD to identify invasive disease due to S.pneumoniae has not been studied in children in sub-Saharan Africa, where high rates of asymptomatic carriage may affect diagnostic accuracy.

Aim:

The overall aim of this study is to evaluate the performance of the ssUAD test to detect pneumococcal carriage, and distinguish it from invasive disease, among children under five years old in Blantyre, Malawi.

Methods:This study will test 350 existing urine samples that have already been collected from children as part of the NP Resistome study (Protocol V 5.0, LSTM reference 24-076), including healthy children in the community, children with pneumonia in the community, and children hospitalised with pneumonia. Participants of the NP Resistome study will be recruited from Ndirande Health Centre (NHC), Gateway Primary Care Centre (GPCC) and Queen Elizabeth Central Hospital (QECH) in Blantyre, Malawi. Aliquots from each urine sample will be tested using the ssUAD in the UK, as the assay is not currently available in Malawi. Urinary detection of pneumococcal serotypes will be compared with both culture-based and metagenomic sequencing results from nasopharyngeal swab samples taken as part of the main study.

DETAILED DESCRIPTION:
Study type: This is a nested case-control sub-study within the multi-site, observational NP Resistome study (COMREC reference P.10/24-1200).

Background:

Pneumococcal pneumonia is a leading cause of morbidity and mortality among children under five, especially in sub-Saharan Africa. Accurate diagnosis remains a challenge due to the need for invasive specimen collection and poor sensitivity of standard culture-based diagnostic tests, particularly after antibiotic use. Serotype-specific urinary antigen detection (ssUAD) offers a promising, non-invasive alternative for serotype surveillance and diagnosis of pneumococcal disease. Serotype-specific identification provided by ssUAD is crucial for monitoring the impact of vaccines and informing public health interventions. The ssUAD test is a Luminex-based urine antigen capture assay developed by the UK Health Security Agency (UKHSA) that targets 24 pneumococcal serotypes, with good sensitivity and specificity among adults with community-acquired pneumonia in the UK. Further investigation is required to determine its ability/utility to identify invasive disease among children, particularly in settings like sub-Saharan Africa, where high rates of asymptomatic carriage may affect diagnostic accuracy.

Broad Objective: To evaluate the performance of the ssUAD test in detecting pneumococcal carriage and distinguishing it from invasive disease among children under five years old in Blantyre, Malawi.

Specific Objectives:

1. To determine the prevalence of serotype-specific pneumococcal antigens in urine among children under five years of age with pneumonia compared to their healthy counterparts.
2. To characterise the association between the detection of serotype-specific antigens in urine and nasopharyngeal pneumococcal carriage among children.
3. To define revised ssUAD thresholds that may distinguish pneumococcal carriage from disease, to support field evaluations and inform diagnostic and surveillance strategies in Malawi and similar settings.

Methodology: We will test 350 existing urine samples that have already been collected from children as part of the NP Resistome study (Protocol v5.0 COMREC reference P.10/24-1200), including healthy children in the community, children with pneumonia in the community, and children hospitalised with pneumonia at the time of recruitment. Participants of the NP Resistome study will be recruited from Ndirande Health Centre (NHC), Gateway Primary Care Centre (GPCC), and Queen Elizabeth Central Hospital(QECH) in Blantyre, Malawi. Urine samples will be aliquoted into 1.8 mL cryotubes and stored at -80°C at Malawi Liverpool Wellcome Research Programme (MLW) laboratory in Malawi. Aliquots from each urine sample will be tested using the ssUAD in the UK, as the assay is not currently available in Malawi. However, we are working towards developing and evaluating the assay locally as part of future implementation efforts. Urinary detection of pneumococcal serotypes will be compared with both culture-based and metagenomic sequencing results from nasopharyngeal swab (NPS) samples taken as part of the main study.

Expected results and dissemination: This sub-study will generate key data on the prevalence of pneumococcal serotype-specific urinary antigens in children with pneumonia and healthy controls. It will improve understanding of ssUAD performance as a surveillance tool in this setting, help distinguish antigenuria due to carriage from disease, and refine diagnostic thresholds for use in high-carriage and disease-burden settings. Study findings will inform surveillance, pneumonia diagnostics, and vaccine impact assessments in LMICs. Results will be shared with COMREC, the Blantyre District Health Office, at scientific conferences, both local and international, and in peer-reviewed publications.

ELIGIBILITY:
Inclusion criteria for healthy children in the community

• Child aged between12-24 months.

Exclusion criteria for healthy children in the community

* Presence of any of the following symptoms: fever, cough, difficulty in breathing or fast breathing.
* Currently taking long-term antibiotic prophylaxis, TB treatment or immunosuppressive medications.
* Diagnosis of an immunosuppressive illness, including HIV infection.
* Hospital admission within the past six months.

Inclusion criteria for children with pneumonia in the community

* Child aged between12-24 months.
* Presence of all of the following symptoms: fever, cough, difficulty in breathing and fast breathing.
* Participant has been prescribed antibiotics for treatment of a lower respiratory tract infection on this presentation.

Exclusion criteria for children with pneumonia in the community

* Severe anaemia, with a recorded haemoglobin level < 70 grams per Litre.
* Currently taking long-term antibiotic prophylaxis, TB treatment or immunosuppressive medications.
* Diagnosis of an immunosuppressive illness, including HIV infection.
* Hospital admission within the past six months.

Inclusion criteria for children hospitalised with pneumonia

* Child aged between 12-24 months.
* Presence of all of the following symptoms: fever, cough, difficulty in breathing and fast breathing.
* Participant has been prescribed antibiotics for treatment of a lower respiratory tract infection on this presentation.

Exclusion criteria for children hospitalised with pneumonia

* Severe anaemia, with a recorded haemoglobin level < 70 grams per Litre.
* Currently taking long-term antibiotic prophylaxis, TB treatment or immunosuppressive medications.
* Diagnosis of an immunosuppressive illness, including HIV infection.
* Hospital admission within the past six months.

Inclusion criteria for children re-hospitalised with pneumonia

* Child aged between12-24 months.
* Presence of all of the following symptoms: fever, cough, difficulty in breathing and fast breathing.
* Participant has been prescribed antibiotics for treatment of a lower respiratory tract infection on this presentation.
* Hospital admission to ANY hospital with a lower respiratory tract infection within the past 3 months.

Exclusion criteria for children re-hospitalised with pneumonia

* Severe anaemia, with a recorded haemoglobin level < 70 grams per Litre.
* Currently taking long-term antibiotic prophylaxis, TB treatment or immunosuppressive medications.
* Diagnosis of an immunosuppressive illness, including HIV infection.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be children aged 12-24 months enrolled in the NP Resistome study (COMREC reference P.10/24-1200) in the following groups;
  * Children hospitalised with pneumonia at Queen Elizabeth Central Hospital.
  * Children with pneumonia treated at Ndirande Health Centre.
  * Healthy children living in Ndirande community.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Serotype specific urinary pneumococcal antigen detection | At the time of recruitment/participant enrolment.
  Serotype-specific urinary pneumococcal antigen detection in urine samples taken at recruitment, using an extended-specificity multiplex urine immunoassay.

SECONDARY OUTCOMES:
Nasopharyngeal pneumococcal carriage | At time of recruitment/enrolment.
  Detection of Streptococcus pneumoniae following culture of nasopharyngeal swab samples on Sheep Blood Agar with 5 µg/mL of Gentamicin (GBA).

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Kwambana-Adams, PhD, Principal Investigator — LSTM

IPD SHARING:
Plan to Share IPD: Yes
Data generated from this sub-study will be shared with collaborators under restricted-access data sharing agreements. All shared datasets will be anonymised and used solely for the purposes outlined in this protocol, in accordance with institutional and ethical guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: Urinary pneumococcal data will be available within 12 months of completion of data collection; approximately October 2027.
  Clinical metadata from the parent study (ISRCTN64027792) will only be available to scientific collaborators, or by application from non-collaborating scientific researchers.
Access Criteria: Anonymised, curated urinary pneumococcal data and clinical metadata will be shared with scientific collaborators. Non-collaborating scientific researchers must submit a formal project proposal for review by investigators to access the data, which if approved, will be released following receipt of a signed data user's agreement setting out roles and responsibilities of data originators and recipients.

DOCUMENTS (1):
  • Study Protocol (2025-08-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT07181200/Prot_000.pdf